CLINICAL TRIAL: NCT00311831
Title: The Implementation of a Gastroenteritis Education Program
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Paediatric Consultants Educational Research Grant (Unknown)
Responsible Party: Principal Investigator, Stephen Freedman, Adjunct Scientist, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1000008727
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Gastroenteritis
Keywords: Pediatrics; Gastroenteritis; Education
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Behavioral: Standard gastroenteritis education
- 2 (Experimental)
  Interventions: Behavioral: Extensive gastroenteritis education

INTERVENTIONS:
Behavioral: Standard gastroenteritis education — Subjects in this arm of the study will receive an educational handout on gastroenteritis education.
  Arms: 1
Behavioral: Extensive gastroenteritis education — Subjects in this arm of the study will receive an gastroenteritis educational handout as well a home visitation from a trained counselor.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the caregivers of children presenting to the emergency department (ED) with acute gastroenteritis who receive extensive gastroenteritis education (standard education plus home nursing visit) will improve their gastroenteritis knowledge more than those who receive standard education (an information sheet) in the emergency department.

DETAILED DESCRIPTION:
Worldwide, diarrhea remains a leading cause of childhood morbidity and mortality, with 2.5 million deaths estimated to occur annually among children < 5 years of age. In the United States, acute gastroenteritis accounts for > 1.5 million outpatient visits, 200,000 hospitalizations and approximately 300 deaths/year. The incidence of diarrhea varies between one and 2.5 episodes per child per year. In Ontario, children account for over 28,000 Emergency Department visits for gastroenteritis annually, and the pediatric admission rate for gastroenteritis remains greater than 400/100,000. In a Toronto based report from 1978, viral gastroenteritis was found as the etiologic agent in the deaths of 21 children over a 5 year period. Over 10% of patients seen at The Hospital for Sick Children ED present with acute gastroenteritis (vomiting, diarrhea or both). Last year over 4500 children with these complaints were seen.

It has been suggested that education can improve caregiver knowledge, beliefs and practices related to gastroenteritis. Children of caregivers who are less knowledgeable about diarrhea, dehydration and oral rehydration have been found to be at increased risk for presenting to a hospital secondary to dehydration.

However, it has been difficult to determine if this will translate into a reduction in non-urgent ED use. Very few studies have evaluated education in the ED. When it has been studied, they have been unsuccessful in altering ED utilization habits. One possible explanation for the lack of success is that some interventions have attempted to teach the parents while they were awaiting discharge. At that point in time, the parents are tired, distracted, and probably anxious to leave, thereby diminishing the effect of the intervention. Furthermore, providing patients with information handouts is not the optimal approach to achieve patient/parent education.

This study will compare two interventions for caregivers of children with gastroenteritis: extensive gastroenteritis education (standard education plus home nursing visit) and standard education in the emergency department(an information sheet). By adding on a home health nurse visit 12 to 36 hours later, we hope to achieve several benefits:

1. Increased parental knowledge regarding gastroenteritis. This includes etiology and prevention, signs and symptoms of dehydration, when to seek care, the appropriate use of oral rehydration solutions, re-feeding, and the role of medications (or lack thereof).
2. Increased parental knowledge will hopefully translate into reduced resource use. This may translate into improved use for other non-acute illnesses such as fever and colds. Improved resource use may include a reduction in ED visits and potentially even primary care provider use.
3. This may also translate into improved patient outcomes by avoiding dehydration, decreasing transmission and seeking medications for the illness. Fewer ED visits may additionally translate into fewer investigations and intravenous requirements.

Thus we will compare improvement in caregiver knowledge of gastroenteritis and dehydration and number of emergency department visits at one year in the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of a child aged 3 months to 4 years of age, presenting to the emergency department with a diagnosis of gastroenteritis, which may be manifested by vomiting, diarrhea, or both
* Age > 16 years
* Ability to speak and read English

Exclusion Criteria:

* Do not live in the metropolitan Toronto area
* Previously enrolled in this trial

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2006-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in parental knowledge as assessed on a gastroenteritis/dehydration questionnaire. | This will be completed on day 1, at 1 month, at 6 months, and at 12 months

SECONDARY OUTCOMES:
Mean score on the caregiver gastroenteritis questionnaire (CGQ) | One year
Number of repeat ED visits for the specific diagnoses of "gastroenteritis", "diarrhea", "vomiting" or "dehydration" | One year

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Freedman, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Freedman SB, Couto M, Spooner L, Haladyn JK. The implementation of a gastroenteritis education program. Am J Emerg Med. 2011 Mar;29(3):271-7. doi: 10.1016/j.ajem.2009.09.032. Epub 2010 Mar 26. PMID 20825796